CLINICAL TRIAL: NCT00086086
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study to Evaluate the Effects of Treatment With 2 Regimens of Subcutaneous Darbepoetin Alfa (Weight-based Dosing and Fixed Dosing) on Hemoglobin Concentration Response in Subjects With Symptomatic CHF and Anaemia
Brief Title: Subcutaneous (SC) Darbepoetin Alfa in Subjects With Symptomatic Congestive Heart Failure (CHF) & Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20020171
Record Dates: First submitted 2004-06-23; First posted 2004-06-24 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Congestive Heart Failure; Anemia
Keywords: Symptomatic Congestive Heart Failure; CHF; Anaemia; Anemia
MeSH Terms: conditions — Heart Failure; Anemia | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin Alfa

SUMMARY:
The purpose of this study is to evaluate whether weight-based or fixed starting doses result in comparable hemoglobin increases and treatment effects in patients with heart failure and anemia.

ELIGIBILITY:
Inclusion Criteria: - Symptomatic CHF for at least 3 months - Reduced left ventricular ejection fraction - Stable heart failure medication - Hemoglobin concentration between 9.0 and 12.5 g/dL Exclusion Criteria: - Hypertension - Unstable angina pectoris or recent myocardial infarction - Likely to receive cardiac transplant - Major organ transplant (e.g., lung, liver, heart) or in renal replacement therapy (e.g., dialysis) - Recent or current treatment for malignancy - Systemic hematologic disease - Anemia due to acute or chronic bleeding - Recent Epogen® or darbepoetin alfa therapy - Recent blood transfusion

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2003-08

PRIMARY OUTCOMES:
Rate of rise of hemoglobin concentration

SECONDARY OUTCOMES:
Change in left ventricular ejection fraction
Change in 6-minute walk distance
NYHA classification
Patient-reported outcomes

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] van Veldhuisen DJ, Dickstein K, Cohen-Solal A, Lok DJ, Wasserman SM, Baker N, Rosser D, Cleland JG, Ponikowski P. Randomized, double-blind, placebo-controlled study to evaluate the effect of two dosing regimens of darbepoetin alfa in patients with heart failure and anaemia. Eur Heart J. 2007 Sep;28(18):2208-16. doi: 10.1093/eurheartj/ehm328. Epub 2007 Aug 6. PMID 17681958
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com